CLINICAL TRIAL: NCT00445783
Title: Melanoma Family Case-Control Study Protocol
Brief Title: Study of Families With Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leeds Cancer Centre at St. James's University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CRUK-LCC-1/3/57; CDR0000532934 (Registry Identifier: PDQ (Physician Data Query)); EU-20704
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-04

CONDITIONS: Melanoma (Skin)
Keywords: lentigo maligna malignant melanoma; stage IV melanoma; acral lentiginous malignant melanoma; nodular malignant melanoma; stage IA melanoma; stage IB melanoma; stage IIA melanoma; stage IIB melanoma; stage IIC melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma
MeSH Terms: conditions — Melanoma | interventions — Gene Expression Profiling; Immunohistochemistry; Restraint, Physical

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: examination
Procedure: mutation carrier screening
Procedure: study of high risk factors

SUMMARY:
RATIONALE: A study that evaluates patients' lifestyle, skin, and blood and tissue samples may help doctors understand the risk factors for melanoma relapse.

PURPOSE: This clinical trial is studying the risk factors for melanoma in families with melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine what lifestyle factors and which genes govern relapse from melanoma.

Secondary

* Compare sun exposure and genes that cause melanoma in patients with melanoma vs healthy participants.
* Assess how unusual moles relate to sun exposure and genes that cause melanoma.

OUTLINE: This is a multicenter, cohort study.

Patients and healthy participants complete lifestyle questionnaires by mail and telephone. Some patients* and healthy participants undergo a skin examination to count moles and classify skin type (e.g., degree of freckling and wrinkling indicative of sun damage).

NOTE: *Patients diagnosed with primary invasive melanoma after September 2005 do not need to consent to a skin examination.

Patients and healthy participants also undergo blood collection for lymphocyte analysis, DNA extraction, and the measurement of minerals, vitamins, and beta carotene. Tissue samples from original diagnosis are examined by immunohistochemistry for gene expression and mutations, including CDKN2A and CDK4.

Patients and healthy participants are followed annually.

Peer reviewed and funded or endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 3,700 patients and healthy participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Newly diagnosed primary invasive melanoma (patient group)

    * Lentigo maligna malignant melanoma allowed
    * Rare variants of melanoma allowed, including any of the following:

      * Acral lentiginous
      * Subungual
      * Ear, nose, and throat
      * Oropharyngeal
      * Perineal
      * Vaginal
      * Vulval
      * Rectal
      * Nodal with no known primary
    * Patients undergoing sentinel node biopsy are eligible
    * No in situ melanoma, melanocytic intraepidermal neoplasia, or ocular melanoma
  * Healthy participant meeting either of the following criteria (control group):

    * Relative of a patient who was diagnosed with melanoma after September 2005
    * Healthy volunteer who is age- and sex-matched for patients who were diagnosed with melanoma before October 2005

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3700 (Estimated)
Dates: Start 2000-07; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Lifestyle factors governing relapse from melanoma
Genes governing relapse from melanoma
Sun exposure and genes that cause melanoma
Unusual moles related to sun exposure and genes that cause melanoma

CONTACTS AND LOCATIONS:
Overall Officials: Julia Newton Bishop, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (1):
- Leeds Cancer Centre at St. James's University Hospital, Leeds, England, United Kingdom